CLINICAL TRIAL: NCT01584128
Title: Use of Structured Non-woven Absorbable Hemostat (or Oxidized Regenerated Cellulose) to Decrease Vaginal Cuff Dehiscence Rate in Laparoscopic Hysterectomy
Brief Title: Oxidized Regenerated Cellulose to Decrease Vaginal Cuff Complications
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 38775EP
Record Dates: First submitted 2012-04-21; First posted 2012-04-24 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Vaginal Cuff Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Oxidized regenerated cellulose: Patients undergoing laparoscopic hysterectomy who have oxidized regenerated cellulose placed at the vaginal cuff at the time of their surgery.

SUMMARY:
The goal of the investigators study is to determine whether the use of oxidized regenerated cellulose reduces the risk of vaginal cuff cellulitis, pelvic abscess, or vaginal cuff dehiscence in patients undergoing laparoscopic hysterectomy. The investigators hypothesize that the use of oxidized regenerated cellulose will reduce the risk of vaginal cuff cellulitis, pelvic abscess, and vaginal cuff dehiscence in patients undergoing laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Structured non-woven absorbable hemostat (or oxidized regenerated cellulose) was designed and marketed for its hemostatic properties. It is used in our practice to achieve hemostasis at the site of the vaginal cuff closure during laparoscopic hysterectomy. While the hemostatic properties of oxidized regenerated cellulose are well known and documented, there is newer research to suggest that oxidized regenerated cellulose may have antimicrobial activity. One In vitro study investigated the antimicrobial activity of oxidized regenerated cellulose products against multiple antibiotic resistant microorganisms and found that the antimicrobial affect of the oxidized regenerated cellulose products was significantly greater than that of the controls. There are a limited number of studies investigating the antimicrobial activity of oxidized regenerated cellulose products in vivo (and none in gynecologic surgery).

ELIGIBILITY:
Inclusion Criteria:

* female, ages 20-80, undergoing laparoscopic hysterectomy

Exclusion Criteria:

* malignant indications for hysterectomy

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women, age 20-80, undergoing laparoscopic hysterectomy
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of vaginal cuff complications | postoperative
  Incidence of vaginal cuff complicationsincluding vaginal cuff dehiscence, vaginal cuff cellulitis, and vaginal cuff abscess

CONTACTS AND LOCATIONS:
Overall Officials: Carrie A Hossler, MD, Principal Investigator — Hershey Medical Center
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States